CLINICAL TRIAL: NCT01642966
Title: Differential Effect of Ticagrelor Versus Prasugrel on the Adenosine-induced Coronary Vasodilatory Responses in Patients With Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor of Cardiology, Director of Cardiology Department, University of Patras
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-12
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Acute Coronary Syndrome
Keywords: ticagrelor; doppler echocardiography
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Active Comparator): Prasugrel 10mg/day for 15 days
  Interventions: Drug: Prasugrel
- Ticagrelor (Experimental): Ticagrelor 90mg twice a day for 15 days
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — Prasugrel 10mg/day for 15 days
  Arms: Prasugrel
Drug: Ticagrelor — Ticagrelor 90mg twice a day for 15 days
  Arms: Ticagrelor

SUMMARY:
This is a prospective, randomized, single-blind, investigator-initiated, crossover study. Patients with Acute Coronary Syndrome (ACS) subjected to percutaneous coronary intervention (PCI), are randomized after informed consent, in a 1:1 ratio to either ticagrelor 90mg x2 or prasugrel 10mg x1 for 15 days. At Day 15± 2 days, coronary diastolic blood flow velocity in left anterior descending artery (LAD) is evaluated at baseline (bCBFV) and under 2 min adenosine infusions (maximal diastolic CBFV- maxCBFV) at gradually increasing doses of 50μg/kg/min, 80μg/kg/min, 110μg/kg/min and 140μg/kg/min with at least 5 min recovery intervals between infusions. A crossover directly to the alternate treatment is performed followed by the same evaluation at Day 30±2 days .

ELIGIBILITY:
Inclusion Criteria:

* Age 18-74 years
* Patients with acute coronary syndrome undergoing PCI with stenting
* Sinus rhythm
* Written informed consent

Exclusion Criteria:

* Known hypersensitivity to prasugrel or ticagrelor
* Requirement for oral anticoagulant prior to the Day 30 visit
* Any previous history of ischemic stroke, intracranial hemorrhage or disease (neoplasm, arteriovenous malformation, aneurysm)
* Any active bleeding or history of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 3 months, other bleeding diathesis, or considered by investigator to be at high risk for bleeding
* Concomitant oral or IV therapy with strong CY P3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazana vir, grapefruit juice N1 L/d), CYP3A substrates with narrow therapeutic indices (cyclosporine, quinidine), or strong CYP3A inducers (rifampin /rifampicin, phenytoin, carbamazepine).
* Increased risk of bradycardiac events.
* Dialysis required.
* Severe uncontrolled chronic obstructive pulmonary disease
* Known severe hepatic impairment
* Pregnancy or breastfeeding
* Left ventricular ejection fraction < 45%, severe left ventricular hypertrophy, diastolic dysfunction, severe valve disease
* Prior myocardial infarction, percutaneous coronary intervention or coronary artery bypass grafting
* Weight < 60 Kg
* Alcohol or narcotics abuse
* Major periprocedural complications: death, cardiogenic shock, stent thrombosis, arrhythmias requiring cardioversion/defibrillation, temporary pacemaker insertion or intravenous antiarrhythmic agents, respiratory failure requiring intubation, retroperitoneal bleeding, major bleeding (need for blood transfusion or drop in haemoglobin post-PCI by ≥ 5 gr/ dl or intracranial bleeding), unsuccessful PCI (residual stenosis > 30% or flow < ΤΙΜΙ 3) or planned staged PCI in the next 5 days after randomization
* Any residual stenosis > 40% in LAD
* Small vessels or diffuse coronary atherosclerosis
* Inability to detect coronary blood flow in LAD

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The area under the curve (AUC) of the maxCBFV (maximal diastolic blood flow velocity in left anterior descending artery)at gradually increasing doses of adenosine | 15 days
  The primary outcome will be assessed 15 days after the onset of each study drug

SECONDARY OUTCOMES:
The ratio of maximal diastolic blood flow velocity in left anterior descending artery/baseline diastolic blood flow velocity in left anterior descending artery for 50μg/kg/min adenosine infusion at the end of treatment periods | 15 days
The ratio of maximal diastolic blood flow velocity in left anterior descending artery/baseline diastolic blood flow velocity in left anterior descending artery for 80μg/kg/min adenosine infusion at the end of treatment periods | 15 days
The ratio of maximal diastolic blood flow velocity in left anterior descending artery/baseline diastolic blood flow velocity in left anterior descending artery for 110μg/kg/min adenosine infusion at the end of treatment periods | 15 days
The ratio of maximal diastolic blood flow velocity in left anterior descending artery/baseline diastolic blood flow velocity in left anterior descending artery for 140μg/kg/min adenosine infusion at the end of treatment periods | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Department Patras University Hospital, Pátrai, Achaia, Greece

REFERENCES:
- [Derived] Alexopoulos D, Moulias A, Koutsogiannis N, Xanthopoulou I, Kakkavas A, Mavronasiou E, Davlouros P, Hahalis G. Differential effect of ticagrelor versus prasugrel on coronary blood flow velocity in patients with non-ST-elevation acute coronary syndrome undergoing percutaneous coronary intervention: an exploratory study. Circ Cardiovasc Interv. 2013 Jun;6(3):277-83. doi: 10.1161/CIRCINTERVENTIONS.113.000293. Epub 2013 Jun 4. PMID 23735473